CLINICAL TRIAL: NCT00263965
Title: A 16-Week Randomized, Double-Blind, Parallel-Group, Multicenter, Placebo- and Active- (Metformin) Controlled Study to Evaluate the Effect on Whole Body Insulin Sensitivity of Tesaglitazar Therapy When Administered to Patients With Type 2 Diabetes
Brief Title: ARAMIS: Actions of tesaglitazaR on fAt Metabolism and Insulin Sensitivity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C09999; EudraCT No 2004-000350-24
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Metformin; Diet

INTERVENTIONS:
Drug: Tesaglitazar
Drug: Metformin
Behavioral: Dietary and lifestyle modification counseling

SUMMARY:
This is a 16-week randomized, double-blind, parallel-group, multi-center, placebo- and active- (metformin 1.5 g) controlled study of tesaglitazar (1 mg) in patients with type 2 diabetes. After a 1-week enrollment period, a 3 week placebo single blind run in period and 1-week placebo single-blind baseline measurement period, the patients will be given the investigational product for 16 weeks in a double blind fashion. Metformin will be titrated up during the first 3 weeks of the double-blind period. The total study duration, including enrollment, run-in, randomized treatment and follow-up, is 29 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are 30-70 years of age
* Female patients: postmenopausal, hysterectomized
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105
Dates: Start 2005-08; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Whole-body insulin sensitivity by assessing the M value during high (80 mU/m2/min) insulin level euglycemic hyperinsulinemic clamp.

SECONDARY OUTCOMES:
Hepatic and peripheral insulin sensitivity by assessing the M value during low (20 mU/m2/min) insulin level euglycemic hyperinsulinemic clamp.
Basal hepatic glucose output measured by dideuterated glucose in the fasting state and during low insulin level clamp.
Plasma profile of glucose, insulin and lipids after a mixed meal
Calculated insulin secretion
Liver oxidation after a mixed meal
Energy expenditure and substrate metabolism by indirect calorimetry
Body composition using DXA-scan, abdominal fat distribution using magnetic resonance imaging, liver fat and muscle fat content using magnetic resonance spectroscopy
Waist and hip circumference
Laboratory efficacy variables (lipids, inflammatory marker and adipose tissue hormones)
Safety and tolerability of tesaglitazar in patients with type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (3):
- Research Site, Helsinki, Finland
- Research Site, Pisa, Italy
- Research Site, Oxford, United Kingdom